CLINICAL TRIAL: NCT07084766
Title: The Variation in Uterine Flexion Angle Before and After Voiding in Parous Women.
Acronym: FLEXIMIX 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 29BRC25.0036; ID RCB (Other: 2025-A00826-43)
Record Dates: First submitted 2025-07-17; First posted 2025-07-25 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Uterine Anteflexion; Parous Women
Keywords: uterine anteflexion; nulliparous women; full bladder; angle of anteflexion or retroflexion of the uterus; ultrasound measurements
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transabdominal ultrasonography (Other): Ultrasound measurements before and after bladder emptying
  Interventions: Procedure: ultrasonography, pelvic

INTERVENTIONS:
Procedure: ultrasonography, pelvic — Ultrasound measurements will be taken before and after bladder emptying. The axes of the uterine body, cervix and vagina will be marked out by tracing the 3 corresponding lines on the image.

SUMMARY:
Intrauterine devices (IUDs) account for approximately 25% of contraceptive methods used in France. However, their insertion can be painful for patients and challenging for practitioners, particularly due to the passage through the cervix and the uterine flexion angle. An interventional study conducted by Cameron in 2013 examined the impact of bladder filling on the ease of IUD insertion. The results did not show a significant benefit, suggesting that a full bladder does not necessarily improve the procedure. An ongoing study, FLEXIMIX, led by the coordinator, explores the variation in the uterine flexion angle based on bladder filling in 250 nulliparous women. Preliminary results indicate a strong influence of bladder filling on the flexion angle. Additionally, the Valsalva maneuver, which involves increasing intra-abdominal pressure by forceful exhalation against a closed glottis, has been shown in two recent studies to facilitate gynecological interventions by improving cervical passage, thereby reducing the need for invasive instruments such as the tenaculum.What happens in parous women and during the Valsalva maneuver remains to be explored.

ELIGIBILITY:
Inclusion Criteria:

* Adult women
* Parous
* Experiencing the need to urinate
* Affiliated with a social security scheme or equivalent

Exclusion Criteria:

* Pregnant women
* Desire for pregnancy with ongoing conception process
* Age > 65 years
* History of hysterectomy
* History of conization
* Childbirth < 6 months
* Irrepressible need to urinate
* Inability or refusal to participate in the study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — have a uterus
Enrollment: 200 (Actual)
Dates: Start 2025-09-25 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Difference between the mean angles of uterine anteflexion and retroflexion with a full and empty bladder in parous women | 1 day
  To determine the difference between the mean angles of uterine anteflexion and retroflexion with a full and empty bladder in parous women

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Brest, Brest, Finistere, France

IPD SHARING:
Plan to Share IPD: Undecided